CLINICAL TRIAL: NCT03877419
Title: Comparison of Different Drilling Speed to Classify Bone Quality by Tactile Sensation on a Saw Bone Model
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201901021RINB
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-01

CONDITIONS: Missing Teeth; Dental Implant
Keywords: dental implant; bone quality; tactile sensation; drilling speed
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of different drilling speed to classify bone quality by tactile sensation on a saw bone model

DETAILED DESCRIPTION:
Bone quality is one of the major factors influencing the dental implant survival rate. Bone quality is believed to have effects on initial implant stability and success of osseointegration. Different implant designs and surgical protocols were developed for improving the survival rate in different bone quality. Although bone quality can be partly diagnosed by radiographic images, lots of experienced surgeons also evaluate bone quality with tactile sensation when they drill the bone. However, variations in evaluation of bone density maybe exist among different surgeons. The drilling speed also may have effect on the outcome of evaluation. For less experienced dentists, it is difficult to diagnose bone quality with tactile sensation in the beginning. The purpose of this study is to find proper drilling speed to classify bone quality by tactile sensation on a saw bone model. Saw bones of variant densities are used as training & testing materials. The proper drilling speed to distinguish different bone quality will be evaluated and offered to junior dentists for better implant treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult dentist, with license no more than 5 years
* No clinical implant surgery experience or with experience less than 10 implants.

Exclusion Criteria:

-Subject who couldn't hold the test procedure

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: junior residents in NTUH
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Units on a Visual Analog Score for bone density | 30 minutes
  the range of the visual analog score was from 0 to 100, 0 indicated drilling into the air, 100 indicated drilling into the hardest jaw bone. The investigators will provide participants several saw bone blocks with different density. Participants needed to answer each bone density of blocks on the scale by drilling feedback sensation after drilling. It's better result that the answers close to the correct bone density of the saw bone blocks.

CONTACTS AND LOCATIONS:
Overall Officials: Tong-Mei Wang, PHD, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan